CLINICAL TRIAL: NCT01049191
Title: Bone Microarchitecture in Women With and Without Fracture
Acronym: mMRI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0177
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-07

CONDITIONS: Osteoporosis; Fracture
Keywords: Osteoporosis; Fracture; microMRI; Bone architecture; Bone matrix; Bone and Bones; Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples are being collected to obtain chemistry panel and test related to skeletal status. These samples will not be retained or stored after these analyses are completed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fracture: Subjects experiencing a prior osteoporotic fracture.
- Control: These will be age and bone density matched controls to the fracture group.

SUMMARY:
Osteoporosis is a common disorder of compromised bone strength causing 40-50% of women and ~25% of men to sustain fragility fractures during their lifetime. The reduction of bone strength in osteoporotic people results from loss of bone density and deterioration of bone quality. Bone quality is a complex amalgamation including macro- and micro-architecture, mineralization, turnover and damage accumulation. Currently, medications to reduce fracture risk are prescribed primarily on the basis of bone mineral density (BMD) measurement. Unfortunately, currently available BMD measurement technologies do not detect the aforementioned properties of bone quality; as such, less than half of individuals who sustain osteoporotic fractures are classified as "osteoporotic" by currently available diagnostic tools. Clearly, measures to enhance identification of those at high fracture risk are needed. High-resolution magnetic resonance imaging (HR-MRI) technology, such as that provided by MicroMRI, Inc., has outstanding potential to be such a tool. Therefore, our long-term goal is to evaluate and optimize the use of HR-MRI in fracture risk prediction; this pilot work is an essential step in attaining this goal.

This research will investigate 72 postmenopausal women with normal or osteopenic BMD by dual-energy x-ray absorptiometry (DXA), 36 with prior low-trauma fractures will be compared with 36 age-, race- and BMD matched women without fracture. We hypothesize that 1.) Women with fractures will have evidence of microarchitectural deterioration on HR-MRI and 2.) Newly developed, more rapid MRI sequences designed at the UW will provide similar trabecular microstructure information more rapidly than the currently used, albeit investigational, technology produced by MicroMRI, Inc.

Our specific aims are to a) Evaluate differences in MicroMRI parameters of trabecular microstructure (bone volume fraction, trabecular thickness, surface/curve ratio and erosion index) between age-, race- and BMD-matched postmenopausal women with and without fracture; b.) Correlate T2* relaxation time (a rapid indirect MRI measure of trabecular density and microstructure) with BMD measured by DXA, and microstructural parameters measured by MicroMRI. As an exploratory aim we will investigate HR-MRI parameters of trabecular microstructure obtained using a newly developed, rapid MRI sequence referred to as IDEAL-FSE with parameters obtained using the currently available MicroMRI, Inc. sequence.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women volunteers age ≥ 50 years
* normal BMD or osteopenia (T-score > -2.5 at the L1-4 spine, proximal femur and 1/3rd radius) by DXA.
* sustained a "fragility" fracture of the spine, hip or wrist, defined as a fracture occurring with everyday activities including a fall from standing height or less.
* Historical radiographic documentation of fracture will be obtained.
* Criteria as defined above without prior fracture, age and bone density matching a participant in the fracture group

Exclusion Criteria:

* metabolic bone disease
* malignancy
* renal failure
* use of medications which alter bone turnover
* diseases/conditions leading to the non-dominant arm disuse
* contraindications to MRI.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seventy-two postmenopausal volunteers age ≥ 50 years will be recruited from existing databases of ~3500 women with expressed interested in research. All will have normal BMD or osteopenia (T-score > -2.5 at the L1-4 spine, proximal femur and 1/3rd radius) by DXA. Thirty-six will have sustained a "fragility" fracture of the spine, hip or wrist, defined as a fracture occurring with everyday activities including a fall from standing height or less. Historical radiographic documentation of fracture will be obtained. Thirty-six women without fracture will serve as age- race- and BMD-matched controls. Age will be matched to within 6 months; BMD in grams/cm2 at the non-dominant ultra-distal radius will be matched to within 5%.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate difference in MicroMRI parameters of trabecular microstructure (bone volume, surface/curve ratio and erosion index) between age-, race- and BMD-matched postmenopausal women with and without fracture. | 18 months

SECONDARY OUTCOMES:
Correlate T2* relaxation time (a rapid indirect MRI measure of trabecular density and microstructure) with BMD measured by DXA, and microstructural parameters measured by MicroMRI. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kijowski, MD, Principal Investigator — University of Wisconsin Department of Radiology; Neil C Binkley, MD, Study Director — University of Wisconsin Osteoporosis Clinical Research Center; Michael J Tuite, MD, Study Director — University of Wisconsin Department of Radiology
Locations (2):
- United States (2):
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - University of Wisconsin Osteoporosis Clinical and Research Program, Madison, Wisconsin